CLINICAL TRIAL: NCT07076810
Title: Morphology of Lumbar Transverse Processes and Relationship With the Success of Lumbar Medial Branch Radiofrequency Ablation in Facet Syndrome
Brief Title: The Relation of the Anatomic Morphology of Lumbar Transverse Processes and the Success Rate of Facet Joint Radiofrequency Denervation
Status: Not yet recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mustafa Kurçaloğlu, Assistant Professor, Ondokuz Mayıs University
Other Study IDs: OMÜ KAEК 2025/252
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Lower Back Pain Chronic
Keywords: lower back pain; radiofrequency; facet joint; transverse process
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group High
  Interventions: Procedure: Lumbar facet joints medial branch nerve radiofrequency ablation

INTERVENTIONS:
Procedure: Lumbar facet joints medial branch nerve radiofrequency ablation — Patients will be positioned prone on the operation table. Intravenous access is opened. Monitorization for vital signs is performed. Light sedation with midazolam is performed. Under fluoroscopic guidance, medial branch nerve of each lumbar facet joint is found by searching the specific response to the stimulations of the radiofrequency needle. When the tip of the radiofrequency needle is close enough to the corresponding medial branch nerve, ablation with 80 degrees Celsius for 90 seconds is performed. Average 6-10 nerves are ablated in each procedure and the average duration of the procedure is 20-60 minutes.
Procedure: Lumbar facet joints medial branch nerve radiofrequency ablation — Patients are positioned prone on the operation table. Intravenous access is opened and monitorization of vital signs is applied. Skin is cleaned by povidone iodine solution. Light sedation is applied by midazolam. Lumbar vertebral region is seen under C-arm fluoroscopic view. Medial branch nerve of the lumbar facet joints is searched by 22 G width, 10-cm length radiofrequency needles. When the needle tip is close enough to the nerve, an 80 Celsius, 90-second radiofrequency ablation is applied. In each procedure, average 5-10 nerves is ablated and the duration of the procedure is 20-60 minutes.

SUMMARY:
Adult patients who were planned for lumbar facet joint medial branch nerve Radiofrequency ablation under fluoroscopic guidance because of facet joint-originated chronic lower back pain will be included in this study. Pain scores (Numerical Rating Scale and Oswestry Disability Index) will be recorded before and one month after the intervention. The morphology of the transverse processes and the facet joints (sizes and angles) will be evaluated using the computer tomography images that patients have in routine examination process. The possible relationship between the success rate of the procedure and the morphology of the transverse processes will be assessed by statistical analysis.

DETAILED DESCRIPTION:
Our study will include patients who are examined at the Ondokuz Mayis University Algology Outpatient Clinic and diagnosed with chronic low back pain originating from the facet joints and deemed suitable for lumbar facet joint medial branch radiofrequency RF ablation (RFA) treatment. The study period will be between August 1, 2025, and June 30, 2026. Those who do not volunteer to participate in the study, those with significant anatomical deformities in the lumbar spine, those unable to answer the study questions, those with a history of lumbar vertebral surgery, and those who are or may be pregnant will be excluded.

Patients' gender, age, body mass index, and the duration of pain will be recorded. Patients' pain intensity will be assessed using the Numerical Rating Scale (NRS) and the Oswestry Disability Index (ODI). The NRS asks patients to rate their pain intensity between 0 and 10. 0 represents no pain, and 10 represents the highest pain they can imagine. Patients' NRS scores and ODI scores at rest and during activity will be recorded before and 1 month after the RFA procedure. A 40% or greater reduction in ODI score will be defined as "significant benefit from the procedure." The angles of the superior articular and transverse processes at the bilateral L1/2, L2/3, L3/4, L4/5, and L5/S1 levels, as well as the angles of the facet joint in the axial plane, will be calculated from Lumbar Spine Computed Tomography images taken during the diagnosis and treatment processes. No additional imaging will be required for this study; the data will be obtained from the patients' previously obtained lumbar spine CT images.

Patients will be divided into two groups for each level: "greater angle" and "lesser angle," based on the angles specified above. Post-procedure pain scores and the rate of significant benefit from the procedure will be compared. Patients will be evaluated one month after the procedure for pain scores and Oswestry Disability Index. Furthermore, a correlation will be investigated between the reduction in pain scores at each level and the specified angles. Statistical analyses of the study will be conducted using Statistical Package for Social Sciences (SPSS) version 26. Data obtained by counting will be expressed as numbers and percentages, and data obtained by measurement will be expressed as mean ± standard deviation. The Student t-test will be used for parameters showing normal distribution in comparisons of descriptive statistical methods and quantitative data, and the Mann-Whitney U test will be used for parameters not showing normal distribution. The chi-square test will be used for comparisons of qualitative data.

The relationship between changes in pain scores and the anatomical angles evaluated in the study will be assessed using the Pearson Correlation Test. A P value of less than 0.05 will be considered statistically significant.

This cross-sectional, observational study will not interfere with the patients' routine treatment protocols.

Sample Size and Statistical Methods: Statistical analyses of the study will be conducted using SPSS (Statistical Package for Social Sciences) version 26. Data obtained by counting will be expressed as numbers and percentages, and data obtained by measurement will be expressed as mean ± standard deviation. The Student t-test will be used for normally distributed parameters when comparing descriptive statistical methods and quantitative data, and the Mann-Whitney U test will be used for non-normally distributed parameters. The chi-square test will be used for comparisons of qualitative data. The relationship between changes in pain scores and the anatomical angles evaluated in the study will be assessed using the Pearson Correlation Test. A P value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar facet joint-originated lower back pain longer then 6 months.

Exclusion Criteria:

* Younger then 18
* Reluctance to participate in the study
* Severe anatomic deformation in lumbar vertebral region
* Presence or suspicion of pregnancy
* Inability to answer the questions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have lumbar facet joint-originated lower back pain for longer than 6 months.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | One month
  Pain assessement tool

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | one month
  A tool for assessment of the severity of low back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The authors of this study may share the participant data when there is a reasonable request.

REFERENCES:
- [Background] Castellvi AE, Goldstein LA, Chan DP. Lumbosacral transitional vertebrae and their relationship with lumbar extradural defects. Spine (Phila Pa 1976). 1984 Jul-Aug;9(5):493-5. doi: 10.1097/00007632-198407000-00014. PMID 6495013
- [Background] Konin GP, Walz DM. Lumbosacral transitional vertebrae: classification, imaging findings, and clinical relevance. AJNR Am J Neuroradiol. 2010 Nov;31(10):1778-86. doi: 10.3174/ajnr.A2036. Epub 2010 Mar 4. PMID 20203111
- [Background] Guan W, Yu W, Lin Q, Zhang Z, Du G, Tian J, Xu Y, Hsieh E. Lumbar Vertebrae Morphological Analysis and an Additional Approach for Vertebrae Identification in Lumbar Spine DXA Images. J Clin Densitom. 2020 Jul-Sep;23(3):395-402. doi: 10.1016/j.jocd.2018.09.004. Epub 2018 Sep 15. PMID 30425005
- [Background] Erken E, Ozer HT, Gulek B, Durgun B. The association between cervical rib and sacralization. Spine (Phila Pa 1976). 2002 Aug 1;27(15):1659-64. doi: 10.1097/00007632-200208010-00013. PMID 12163729